CLINICAL TRIAL: NCT07156357
Title: sEMG Assessment of Swallowing and Bolus Preparation
Brief Title: Surface EMG Testing on Swallowing in EoE Patients
Acronym: sEMG
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karthik Ravi, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 24-009832
Record Dates: First submitted 2025-08-15; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Subjects who can swallow normally
  Interventions: Diagnostic Test: Surface Electromyography; Diagnostic Test: Fiberoptic Endoscopic Evaluation of Swallowing
- Eosinophilic Esophagitis: Subjects with Eosinophilic Esophagitis
  Interventions: Diagnostic Test: Surface Electromyography; Diagnostic Test: Fiberoptic Endoscopic Evaluation of Swallowing

INTERVENTIONS:
Diagnostic Test: Surface Electromyography — Tests performed to evaluate swallowing function
Diagnostic Test: Fiberoptic Endoscopic Evaluation of Swallowing — Assessment of swallowing function

SUMMARY:
Evaluating swallowing food with surface electromyography (EMG) machine in patients with Eosinophilic Esophagitis

DETAILED DESCRIPTION:
Evaluating surface electromyography (sEMG) assessment of swallowing and bolus preparation in patients with Eosinophilic Esophagitis (EoE).

ELIGIBILITY:
Inclusion Criteria:

* Controls

  * Normal video swallow or score of 0 for dysphagia on ESSAI questionnaire
  * absence of dysphagia
  * age >18 EoE participants
  * Documentation of EoE diagnosis by histologic criteria,
  * >15 eos/hpf on most recent esophageal biopsy
  * age >18

Exclusion Criteria:

* Abnormal baseline video swallow
* lack of MSK coordination to eat test meal
* underlying neuromuscular disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit patients with EoE seen in the esophageal clinic. Controls will be recruited by monitoring for patients that present for video swallow with speech language pathology and have a normal video swallow.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Preparatory phase time | Through study completion an average of 2 days
  Comparison of preparatory phase between cohorts

SECONDARY OUTCOMES:
Time difference in swallow initiation | Through study completion an average of 2 days
  Time difference in swallow initiation between fiberoptic endoscopic evaluation of swallowing (FEES) vs sEMG

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ravi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No